CLINICAL TRIAL: NCT06410404
Title: Dexmeditomedine as an Adjuvant to Levobupivacaine in Transversus Thoracis Plane Block on the Management of Post-sternotomy Pain in Open-heart Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed wahby Shamsedine, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: post-sternotomy pain control
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Levobupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine group (Active Comparator): * Patients in this group shall receive levobupivacaine alone.
  * Transversus thoracic plane block will be carried out with the patient lying in the supine position. After skin disinfection, a high frequency linear ultrasound probe will be applied parallel to and between the 4th and 5th ribs connecting at the sternum. Then, 15 ml of levobupivacaine 0.25% will be injected between the transversus thoracic muscle and the internal intercosatal muscle.
  Interventions: Procedure: transversus thoracis plane block; Drug: Levobupivacaine
- Combined levobupivacaine, and dexmeditomedine group (Active Comparator): * Patients in this group shall receive levobupivaciane in addition to dexmeditomedine as an adjuvant.
  * Transversus thoracic plane block will be carried out with the patient lying in the supine position. After skin disinfection, a high frequency linear ultrasound probe will be applied parallel to and between the 4th and 5th ribs connecting at the sternum. Then, 15 ml of levobupivacaine 0.25%, together with dexmeditomedine in a dose of 1 ug/kg will be injected between the transversus thoracic muscle and the internal intercosatal muscle.
  Interventions: Procedure: transversus thoracis plane block; Drug: Dexmedetomidine; Drug: Levobupivacaine

INTERVENTIONS:
Procedure: transversus thoracis plane block — with the patient lying in the supine position. After skin disinfection, a high frequency linear ultrasound probe will be applied parallel to and between the 4th and 5th ribs connecting at the sternum. Then, different drugs according to the different groups will be injected between the transversus thoracic muscle and the internal intercosatal muscle.
  Other Names: TTPB
Drug: Dexmedetomidine — the dexmeditomedine group shall undergo bilateral transversus thoracis plane block with 15 ml of 25% levobupivacaine, and 0.05 ug/kg dexmeditomedine on each side of the sternum
  Arms: Combined levobupivacaine, and dexmeditomedine group
Drug: Levobupivacaine — A local anesthetic that will be instilled in the transversus thoracic plane in a dose of 15 ml of a 25% concentration on both sides of the sternum in both groups

SUMMARY:
the study is to assess the efficacy of dexmeditomedine as an adjuvant to the local anaesthetic levobupivacaine in transversus thoracis plane block given bilaterally on the management of post-sternotomy pain.

DETAILED DESCRIPTION:
the patients will fall into one of two groups using an online randomizer. this study is an assessor-blinded interventional controlled study. the first group will recieve transversus thoracis plane block bilaterally where 15 ml of 0.25% levobupivacaine will be given. and the other group shall also undergo a bilateral transversus thoracis plane block with 15 ml 0.25% levobupivacaine and 0.05 ug/kg dexmeditomedine on each side. the primary aim of the study is the 24 hour post-operative morphine consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 20 years old.
* ASA II to III patients undergoing elective cardiac surgery via a median sternotomy

Exclusion Criteria:

* Patient's refusal.
* Known contraindications to regional blocks, including local skin infections,and coagulopathy.
* Allergies to the local anaesthetics used.
* Patients undergoing complex cardiac procedures.
* Patients with severe chronic obstructive pulmonary disease.
* Patients unable to communicate.
* Patients with chronic pain.
* Patients with severe pulmonary hypertension.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Total post-operative morphine consumption. | 24 hours post-operative
  If the patient experiences a pain of > 4, he will be given morphine intravenously in a dose of 0.05 mg/kg IV by a blinded assessor, aiming for a pain score of ≤ 4. The total morphine dose for the post-operative 24 hours will be compared between the case and control group, to determine which technique provided more analgesia.

SECONDARY OUTCOMES:
Post-operative pain score | 24 hours post-operative
  VAS (Visual Analogue Scale, 0-10; where 0 = no pain, and 10 = worst imaginable pain) will be assessed at rest, preoperatively, half an hour after extubation, and at 4th, 8th, 12th, 16th, 20th, and 24th hours post operatively. Moreover, VAS will also be assessed at 12th and 24 hours post-operatively while coughing.
Time till request of first analgesia. | 24 hours post-operative
  comparison of the time till request of first analgesia difference between the two groups, shall give us a clue to the effect of demeditomedine on the duration of the pain controlling effect of the used block.
Intensive Care Unit (ICU) stay length. | 4 days
  time till discharge from the ICU
Complications of the interventional block | 24 hours post-operative
  * Pneumothorax.
  * Hemothorax.
  * Local anaesthetic systemic toxicity.
  * Intravascular injection.
  * Allergy to the local anaesthetic used.
  * Infection.
  * Hematoma.
  * Neural injury.
  * Damage to internal thoracic artery.

IPD SHARING:
Plan to Share IPD: Undecided
the decision shall be taken at the end of the study. I anticipate that it is going to be a "yes".

REFERENCES:
- [Background] Mazzeffi M, Khelemsky Y. Poststernotomy pain: a clinical review. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1163-78. doi: 10.1053/j.jvca.2011.08.001. Epub 2011 Sep 29. No abstract available. PMID 21955825
- [Background] El-Ansary D, LaPier TK, Adams J, Gach R, Triano S, Katijjahbe MA, Hirschhorn AD, Mungovan SF, Lotshaw A, Cahalin LP. An Evidence-Based Perspective on Movement and Activity Following Median Sternotomy. Phys Ther. 2019 Dec 16;99(12):1587-1601. doi: 10.1093/ptj/pzz126. PMID 31504913
- [Background] Liu SS, Wu CL. Effect of postoperative analgesia on major postoperative complications: a systematic update of the evidence. Anesth Analg. 2007 Mar;104(3):689-702. doi: 10.1213/01.ane.0000255040.71600.41. PMID 17312231
- [Background] Popping DM, Elia N, Marret E, Remy C, Tramer MR. Protective effects of epidural analgesia on pulmonary complications after abdominal and thoracic surgery: a meta-analysis. Arch Surg. 2008 Oct;143(10):990-9; discussion 1000. doi: 10.1001/archsurg.143.10.990. PMID 18936379
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Moon MH, Kang JK, Kim HW, Jo KH, Choi SH, Song H. Pain after median sternotomy: collateral damage or mitigatable byproduct? Thorac Cardiovasc Surg. 2013 Apr;61(3):194-201. doi: 10.1055/s-0032-1311540. Epub 2012 Nov 6. PMID 23132359
- [Background] Huang AP, Sakata RK. [Pain after sternotomy - review]. Rev Bras Anestesiol. 2016 Jul-Aug;66(4):395-401. doi: 10.1016/j.bjan.2014.09.003. Epub 2015 Mar 18. Portuguese. PMID 25796483
- [Background] Raj N. Regional anesthesia for sternotomy and bypass-Beyond the epidural. Paediatr Anaesth. 2019 May;29(5):519-529. doi: 10.1111/pan.13626. PMID 30861264
- [Background] Ueshima H, Kitamura A. Blocking of Multiple Anterior Branches of Intercostal Nerves (Th2-6) Using a Transversus Thoracic Muscle Plane Block. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):388. doi: 10.1097/AAP.0000000000000245. No abstract available. PMID 26079353
- [Background] Walian A, Magoon R, Shri I, Kashav RC. Transversus Thoracic Muscle Plane Block for Attenuating the Haemodynamic Response to Median Sternotomy: A Case Series. Turk J Anaesthesiol Reanim. 2022 Dec;50(6):449-453. doi: 10.5152/TJAR.2022.21196. PMID 36511495
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179
- [Background] Shokri H, Ali I, Kasem AA. Evaluation of the Analgesic Efficacy of Bilateral Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Post-Sternotomy Pain: A Randomized Controlled Trial. Local Reg Anesth. 2021 Nov 12;14:145-152. doi: 10.2147/LRA.S338685. eCollection 2021. PMID 34803399
- [Background] Chen Z, Liu Z, Feng C, Jin Y, Zhao X. Dexmedetomidine as an Adjuvant in Peripheral Nerve Block. Drug Des Devel Ther. 2023 May 17;17:1463-1484. doi: 10.2147/DDDT.S405294. eCollection 2023. PMID 37220544
- See also: Ball M, Falkson SR, Fakoya AO, et al. Anatomy, Angle of Louis. [Updated 2023 Dec 10]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2024 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK459336/ — https://www.ncbi.nlm.nih.gov/books/NBK459336/